CLINICAL TRIAL: NCT04600050
Title: Effect of Eccentric Contraction-based Resistance Exercise on Functional Recovery in Chronic Stroke Patients
Brief Title: Eccentric Contraction-based Resistance Exercise for Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Jae-Young Lim, Professor, Department of Rehabilitation Medicine, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NRCRSP-EX20010
Record Dates: First submitted 2020-09-15; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Stroke
Keywords: Eccentric exercise; Stroke; Physical function; Muscle function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: stroke patients with education (Active Comparator)
  Interventions: Other: usual care and exercise education
- Experimental: stroke patients with exercise (Experimental)
  Interventions: Other: Eccentric exercise

INTERVENTIONS:
Other: usual care and exercise education — Provide exercise training materials after the education of exercise and health to enable home-based exercise
  Arms: Control group: stroke patients with education
Other: Eccentric exercise — Under the face-to-face supervisor, the eccentric exercise using a flywheel, and the self-directed home-based eccentric overload exercise using an elastic band are performed.
  Arms: Experimental: stroke patients with exercise

SUMMARY:
The purpose of this study is to develop an evidence-based rehabilitation treatment method suitable for recovery and improvement of physical function in chronic stroke patients using an eccentric overload flywheel device. Participants are disabled with chronic stroke (ischemic and hemorrhagic cerebral hemorrhage) over 50 years of age, who can communicate with a Korean simple mental state test (MMSE-K) of 24 points or higher, and whose functional gait score is 3-5 points. The investigators will enroll 40 participants and randomly assign them to either the control (Con, n=20) or the exercise (Ex, n=20) group. The investigators will verify the effectiveness of the exercise program through the evaluation of changes in muscle and physical function before and after intervention in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with disabilities 50 years of age or older who have been diagnosed with a stroke (ischemic and hemorrhagic cerebral hemorrhage) for at least one year
* Patients can communicate with a Korean simple mental state test (MMSE-K) of 24 points or higher
* Patients have a functional ambulation category (FAC) score of 3 to 5

Exclusion Criteria:

* Patients with brain lesions and quadriplegia excluding stroke
* Patients with uncontrolled hypertension with limited exercise intervention
* Patients diagnosed with angina
* Patients with congestive heart failure (CHF)
* Patients with upper/lower extremity fracture within 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Isokinetic knee extensor strength | Change from Baseline muscle function at 8 weeks of intervention.
  Evaluation of change from baseline isokinetic knee extensor strength to 8 weeks after the initial assessment. Isokinetic knee extensor strength is measured in peak torque (Nm) achieved on an isokinetic dynamometer (BTE Primus, BTE tech, MD, USA) at 60° per second.
Short physical performance battery (SPPB) scores | Change from Baseline physical function at 8 weeks of intervention.
  Evaluation of change from baseline SPPB score to 8 weeks after the initial assessment. The SPPB is a group of measures that combine the results of the gait speed, timed chair stand and balance tests. For the static standing balance test, participants were asked to stand in side-by-side, semi-tandem and tandem positions, and maintain each position for 10 s. For the gait speed test, participants were asked to walk along a 4-m distance at their normal walking speed. For the repeated chair rise test, participants were asked to fold their arms across their chest and stand up from a sitting position five times consecutively as quickly as possible. Performance scores for each SPPB individual test and a summary score aggregating the individual tests were calculated as per standard SPPB protocol (range 0-12). The scores range from 0 (worst performance) to 12 (best performance).

SECONDARY OUTCOMES:
Hand grip strength | Change from Baseline physical function at 8 weeks of intervention
  Evaluation of change from baseline hand grip strength to 8 weeks after the initial assessment. Participants are tested while they were seated, their arms are against their sides, their elbows are flexed 90 degrees. Hand grip strength is measured in kilograms (kg) using a hand-grip dynamometer (Takei 5401, Tokyo, Japan). The maximum value from either hand is used for analysis.
Isotonic knee power | Change from Baseline physical function at 8 weeks of intervention
  Evaluation of change from baseline isotonic knee power to 8 weeks after the initial assessment. knee extension and flexion were performed as quickly as possible during a period of 10 seconds and is measured in watts.
Isometric knee strength | Change from Baseline physical function at 8 weeks of intervention
  Evaluation of change from baseline isometric knee strength to 8 weeks after the initial assessment. Isometric knee strength was measured in Newton-meters (Nm) using a baltimore therapeutic equipment (BTE) Primus RS (BTE Tech., Hanover, MD, USA). The participants were asked to sit on the treatment chair and a standard stabilization strap was placed on the upper ankle. The knee was kept at 90 degree flexion, and the foot was positioned in dorsi-flexion.
Isokinetic knee extensor eccentric strength | Change from Baseline muscle function at 8 weeks of intervention.
  Evaluation of change from baseline isokinetic knee extensor eccentric strength to 8 weeks after the initial assessment. Isokinetic knee extensor eccentric strength is measured in peak torque (Nm) achieved on an isokinetic dynamometer (BTE Primus, BTE tech, MD, USA) at 30° per second.
Timed up and go | Change from Baseline physical function at 8 weeks of intervention.
  Evaluation of change from baseline timed up and go to 8 weeks after the initial assessment. Participants sat on a chair and measured the time (second) that it took the participants to stand up, walk 3 m as quickly and safely as possible, turn around at a marked line on the floor, walk back, and sit down.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anker SD, von Haehling S. Efforts begin to sprout: publications in JCSM on cachexia, sarcopenia and muscle wasting receive attention. J Cachexia Sarcopenia Muscle. 2014 Sep;5(3):171-6. doi: 10.1007/s13539-014-0158-6. Epub 2014 Sep 6. No abstract available. PMID 25192875
- [Background] Arvanitidis A, Henriksen K, Karsdal MA, Nedergaard A. Neo-epitope Peptides as Biomarkers of Disease Progression for Muscular Dystrophies and Other Myopathies. J Neuromuscul Dis. 2016 Aug 30;3(3):333-346. doi: 10.3233/JND-160150. PMID 27854226
- [Background] Chang TF, Liou TH, Chen CH, Huang YC, Chang KH. Effects of elastic-band exercise on lower-extremity function among female patients with osteoarthritis of the knee. Disabil Rehabil. 2012;34(20):1727-35. doi: 10.3109/09638288.2012.660598. Epub 2012 Mar 8. PMID 22397710
- [Background] Choi SJ, Lim JY, Nibaldi EG, Phillips EM, Frontera WR, Fielding RA, Widrick JJ. Eccentric contraction-induced injury to type I, IIa, and IIa/IIx muscle fibers of elderly adults. Age (Dordr). 2012 Feb;34(1):215-26. doi: 10.1007/s11357-011-9228-2. Epub 2011 Mar 24. PMID 21431924
- [Background] Roig M, Macintyre DL, Eng JJ, Narici MV, Maganaris CN, Reid WD. Preservation of eccentric strength in older adults: Evidence, mechanisms and implications for training and rehabilitation. Exp Gerontol. 2010 Jun;45(6):400-9. doi: 10.1016/j.exger.2010.03.008. Epub 2010 Mar 18. PMID 20303404
- [Background] Lim JY. Therapeutic potential of eccentric exercises for age-related muscle atrophy. Integr Med Res. 2016 Sep;5(3):176-181. doi: 10.1016/j.imr.2016.06.003. Epub 2016 Jun 18. PMID 28462115
- [Background] Kim KE, Jang SN, Lim S, Park YJ, Paik NJ, Kim KW, Jang HC, Lim JY. Relationship between muscle mass and physical performance: is it the same in older adults with weak muscle strength? Age Ageing. 2012 Nov;41(6):799-803. doi: 10.1093/ageing/afs115. Epub 2012 Aug 21. PMID 22910301
- [Background] Kim YH, Kim KI, Paik NJ, Kim KW, Jang HC, Lim JY. Muscle strength: A better index of low physical performance than muscle mass in older adults. Geriatr Gerontol Int. 2016 May;16(5):577-85. doi: 10.1111/ggi.12514. Epub 2015 May 28. PMID 26017097
- [Derived] Kim Y, Oh S, Kim DY, Lim JY. Effects of eccentric contraction-based resistance exercise on physical performance in chronic stroke patients: A randomized controlled trial. Medicine (Baltimore). 2025 Aug 8;104(32):e43491. doi: 10.1097/MD.0000000000043491. PMID 40797445